CLINICAL TRIAL: NCT05471622
Title: Study of Home-Embedded Palliative Care for Hemodialysis-Dependent End-Stage Renal Disease
Acronym: SHEPHERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Scott Halpern, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 851328
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: End-Stage Renal Disease
Keywords: palliative; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The lead case manager and covering provider on the inpatient care team for participants in this group will receive a message from the research team identifying their patient as appropriate for home palliative care and will be asked to refer their patient for these services.
  Interventions: Behavioral: Nudge for PHPC Referral
- Usual Care (No Intervention): Participants in this group will receive usual care upon discharge from the hospital. Their clinical team will not be notified that they are appropriate for home palliative care services, but they may still be referred for those services if their clinicians feel their patient will benefit.

INTERVENTIONS:
Behavioral: Nudge for PHPC Referral — The case manager and covering providers for inpatients who have been identified according to the study's inclusion criteria as appropriate for Penn Home Palliative Care (PHPC) upon hospital discharge will be asked to refer their patient for these home palliative care services.
  Arms: Intervention

SUMMARY:
Home palliative care needs are often under-recognized in patients with End-Stage Renal Disease (ESRD). This pilot study is designed to evaluate the feasibility and acceptability of an initiative to enhance referrals to Penn Home Palliative Care compared with usual care among hemodialysis-dependent ESRD patients admitted to a Penn hospital. Results will inform a future pragmatic trial comparing the effectiveness of home palliative care compared with usual care among ESRD patients. Evaluating the effectiveness of home palliative care services is critical to determine whether increasing access to these services would improve patient-centered outcomes for these high-need patients.

ELIGIBILITY:
Inclusion Criteria:

* Be an adult (18 years of age or older) hospitalized at one of two study hospitals
* Digital signature of ESRD (N18.6) within the last 12 months with an inpatient hemodialysis order
* Patient resides in the five-county area surrounding Philadelphia which is served by the Penn Home Palliative Care services.
* Appropriate for home palliative care, defined as:

  (i) Existing home care eligibility/referral for home care OR (ii) Severe protein malnutrition (E43, E44) OR (iii) Non-ambulatory status determined by a flowsheet completed by nursing on hospital admission with three ambulatory options: (1) non-ambulatory, (2) ambulates with assistance, or (3) ambulates independently. If this information is missing from the electronic health record, the determination will be made using one of the three following options: (1) overall prior home mobility assessment "complete dependence on all aspects," or (2) ambulation or functional transfers domains indicate "dependent," or (3) wheelchair mobility domain was completed (with any non-null/non-empty value).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Rate of Home Palliative Care Receipt | Baseline - 45 days
  Receipt of home palliative care will be defined as at least one home palliative care visit within 45 days after hospital discharge, determined via electronic health record review.

SECONDARY OUTCOMES:
Follow-up Home Palliative Care Visits | Baseline - 180 days
  The total number of home palliative care visits during the 180-day follow-up period after hospital discharge will be assessed using the electronic health record.
Mortality | Baseline - 180 days
  Mortality rates will be assessed using the electronic health record after the 180-day follow-up period.
Hospital-free days | Baseline - 180 days
  The number of hospital-free days during the 180-day follow-up period will be assessed using the electronic health record and administrative data for the tri-state area.
Acceptability of home palliative care referral among clinician stakeholders | Baseline - 180 days
  Acceptability of home palliative care referral among clinician stakeholders will be measured via survey and focus group questions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No